CLINICAL TRIAL: NCT01423357
Title: Targeting Interventions at Venues Where Risk of HIV Transmission is High
Acronym: PLACE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zambia (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Principal Investigator, Ingvild Fossgard Sandoy, Researcher, University of Bergen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PLACE
Record Dates: First submitted 2011-08-23; First posted 2011-08-25 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: HIV
Keywords: HIV prevention; condom distribution; youth peer education; high risk places; condom use; prevention through increased condom use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Condom distribution and peer education (Experimental): Youth peer educators distribute condoms and conduct condom demonstration in venues where people meet new sexual partners, i.e. bars, night clubs, sherbeens, guest houses
  Interventions: Other: Condom distribution and peer education
- Business as usual (No Intervention)

INTERVENTIONS:
Other: Condom distribution and peer education — Condom distribution and condom demonstrations by youth peer educators at least twice a week
  Arms: Condom distribution and peer education

SUMMARY:
The aim of this study is to investigate whether distribution of condoms and condom demonstrations by youth peer educators in venues where people meet new sexual partners in Livingstone, Zambia, leads to increased condom use among guests socializing in these venues.

DETAILED DESCRIPTION:
In countries where the HIV prevalence is high, focusing on high risk places such as venues where people meet new sexual partners is probably more effective in reducing the transmission rate of HIV than targeting interventions just at perceived high risk groups. A survey conducted in 2005 in places where people met new sexual partners in Livingstone found that guests socializing there were engaging in high risk sex, but condoms were not always available in the venues. In this intervention study, youth peer educators will distribute condoms and demonstrate condom use in venues where people meet new sexual partners. After the intervention has run for a year, condom use among guests socializing in such venues in the intervention township will be compared with condom use among people socializing in similar venues in a comparison township.

ELIGIBILITY:
Inclusion Criteria:

* Socializing in a venue where people are said to be meeting new sexual partners
* Age 18 years and above

Exclusion Criteria:

* Too drunk to give sensible answers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2009-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Condom use with last sexual partner met in this venue | in post-intervention survey (1 year after start of intervention)
  Guests socializing in venues where people meet new sexual partners are asked about condom use with the last sexual partner met in the venue where interview conducted

SECONDARY OUTCOMES:
Condom availability in the last 12 months in venues where people meet new sexual partners | in post-intervention survey (1 year after start of intervention)
  One person representing each venue included in the survey is asked about the availability of condoms in the venue in the last 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles C Michelo, MD, MPH, PhD, Study Director — University of Zambia; Cosmas M Zyaambo, MD, MPhil, Principal Investigator — University of Zambia; Knut M Fylkesnes, DMD. DrPhilos, Study Chair — University of Bergen
Locations (2):
- Zambia (2):
  - Dambwa, Livingstone
  - Maramba, Livingstone

REFERENCES:
- [Background] Sandoy IF, Siziya S, Fylkesnes K. Lost opportunities in HIV prevention: programmes miss places where exposures are highest. BMC Public Health. 2008 Jan 24;8:31. doi: 10.1186/1471-2458-8-31. PMID 18218124
- [Derived] Sandoy IF, Zyaambo C, Michelo C, Fylkesnes K. Targeting condom distribution at high risk places increases condom utilization-evidence from an intervention study in Livingstone, Zambia. BMC Public Health. 2012 Jan 5;12:10. doi: 10.1186/1471-2458-12-10. PMID 22221738